CLINICAL TRIAL: NCT02457585
Title: Anti-tumor Necrosis Factor Therapy Effect on Takayasu Arteritis
Brief Title: Clinical Study of Anti-tumor Necrosis Factor Therapy in Patients With Takayasu Arteritis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1312-079-541
Record Dates: First submitted 2015-05-18; First posted 2015-05-29 (Estimated); Last update posted 2017-05-15 (Actual); Status verified 2017-03

CONDITIONS: Takayasu's Arteritis
MeSH Terms: conditions — Takayasu Arteritis | interventions — Infliximab; CT-P13

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- experimental group (Experimental): anti Tumor necrosis factor treatment group : treatment with remicade 5mg/kg as scheduled (0, 2, 6, 14, 22, 30, 38, 46, 54weeks).
  evaluation of response at 30weeks by PET CT, acute phase reactants, symptom
  No placebo group
  Interventions: Drug: remicade (anti tumor necrosis factor inhibitor)

INTERVENTIONS:
Drug: remicade (anti tumor necrosis factor inhibitor) — single arm:remicade treatment group
  Other Names: remsima

SUMMARY:
Clinical study of anti-tumor necrosis factor therapy in patients with Takayasu arteritis.

This study is single arm (anti Tumor necrosis factor therapy only) clinical trial. Enrolled patients will be 11

DETAILED DESCRIPTION:
Clinical study of anti-tumor necrosis factor therapy in patients with Takayasu arteritis.

This study is single arm (anti Tumor necrosis factor therapy only) clinical trial. Enrolled patients will be 11 patients with active takayasu's arteritis

ELIGIBILITY:
Inclusion Criteria:

* active takayasu's arteritis

Exclusion Criteria:

* active Tuberculosis
* Liver function abnormality
* heart failure ( New York Heart Association III - IV)
* patients were not consented

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Estimated)
Dates: Start 2015-03; Primary Completion 2017-08 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
remission induction at 30 weeks | 30 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yeong Wook Song, MD,PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Park EH, Lee EY, Lee YJ, Ha YJ, Yoo WH, Choi BY, Paeng JC, Suh HY, Song YW. Infliximab biosimilar CT-P13 therapy in patients with Takayasu arteritis with low dose of glucocorticoids: a prospective single-arm study. Rheumatol Int. 2018 Dec;38(12):2233-2242. doi: 10.1007/s00296-018-4159-1. Epub 2018 Sep 18. PMID 30229280